CLINICAL TRIAL: NCT01414660
Title: Adipocytes, Insulin Resistance and Immunity: Evolution of Interleukin 7, Fat Mass and Metabolic Profile Before and After Transplantation
Brief Title: Evolution of Interleukin 7, Fat Mass and Metabolic Profile Before and After Transplantation
Acronym: IL-7tran
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_09/0940; 2009-A01169-48 (Other: ID-RCB number, ANSM); B91413-80 (Other: AFSSAPS); PHRC 2009/API (Other: DHOS)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Immunodeficiency Secondary to Organ Transplantation
Keywords: interleukin 7; transplantation; liver; kidney; islet; diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — wholeblood and tissue bank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- islet: type 1 diabetic patients undergoing islet transplantation
  Interventions: Procedure: transplantation
- liver: non diabetic patients undergoing a liver transplantation
  Interventions: Procedure: transplantation
- kidney: non diabetic patients undergoing a kidney transplantation
  Interventions: Procedure: transplantation

INTERVENTIONS:
Procedure: transplantation — transplantation of islet, kidney or liver

SUMMARY:
Three different white adipose tissue-related disorders, whether due to its excess (obesity), absence (lipoatrophies) or aberrant distribution (lipodystrophies), are paradoxically able to induce metabolic insulin resistance syndrome. The respective roles played by quantitative and qualitative anomalies of adipose tissue, gluco- and lipo-toxicity, liver and muscle insulin resistance, low-grade fat inflammation and immune alterations are not yet perfectly understood. In contrast to most organ transplantations that are often complicated by post-transplantation diabetes, diabetes cell therapy is associated with body weight loss, which is possibly related to the antiadipogenic effects of mTOR inhibitors (rapamycin or sirolimus). The aim of this study is thus to determine and monitor blood interleukin-7 and other cytokine levels; metabolic parameters; and fat mass distribution with DEXA and RMN, before and after a immunosuppressive regimen in patients receiving different kinds of transplantation (liver, kidney or islets) with normal weight and no type 2 diabetes before transplantation. In these patients, blood samples will be taken before and after transplantation, as will adipose tissue during the transplantation surgery, in order to constitute a plasma serum, gene and tissue bank for improving our knowledge of disorders linking fat mass, insulin resistance and immunity, especially post-transplantation diabetes.

DETAILED DESCRIPTION:
Rationale: Due to their ability to store fatty acids and to secrete numerous pro-inflammatory cytokines, adipocytes appear to be key cells in the regulation of energy metabolism and immune response. Moreover, it has been recently shown that adipocytes play a role in the recruitment of cells involved in innate and adaptive immunity in adipose tissue.

White adipose tissue-related diseases are numerous, whether from its excess (obesity), or its complete (lipoatrophies) or partial absence (lipodystrophies); these 3 different disorders are paradoxically able to induce metabolic insulin resistance syndrome.

Among the involved cytokines, interleukin-7 (IL-7), mostly known for its immune functions, also participates in the quantitative and qualitative balance of fat mass. Thus, IL-7 over-expression in animal models induces a lipodystrophic syndrome with insulin resistance, whereas in humans a preliminary study shows that LMNA-linked lipodystrophies are associated with an increase of blood IL-7 levels. IL-7 also participates in reactivation of autoimmunity in patients with autoimmune type 1 after islet transplantation.

Otherwise, mammalian target of rapamycin (mTOR) inhibitors have immunosuppressive, metabolic and anti-tumoral properties through different signaling pathways. Rapamycin (or sirolimus) (Rapamune®), an mTOR inhibitor used in islet transplantation, has much greater ability to inhibit adipocyte differentiation and to modulate ß cell function according to the energetic status. In contrast to most organ transplantation, diabetes cell therapy is associated with body weight loss, which is possibly related to the antiadipogenic effects of mTOR inhibitors; the specific role that this plays on the prognostic factors of islet transplantation remains to be determined. Conversely, organ transplantation is usually associated with weight gain, which is involved in the genesis of post-transplantation diabetes, AKA new-onset diabetes after transplantation (NODAT), and long-term vascular complications of transplantation. Adipose tissue redistribution has not yet been studied in patients after transplantation.

The aim of this study is thus to determine blood IL-7 and other cytokine levels; metabolic parameters; and fat mass distribution before and after a immunosuppressive regimen in patients receiving different kinds of transplantation (liver, kidney or islets) with normal weight and no type 2 diabetes before transplantation. In these patients, blood samples will be taken before and after transplantation, as will adipose tissue during the transplantation surgery, in order to constitute a plasma, serum, gene and tissue bank for determining the mechanisms linking fat mass, insulin resistance and immunity, both ex vivo and in vitro.

Patients: The included patients are normal-weight subjects enlisted for liver, kidney or islet transplantation, with no type 2 diabetes (for liver and kidney transplantation).

Methods: Blood IL-7 levels, other immune and/or pro-inflammatory cytokines, lymphocyte immunophenotype, metabolic parameters, and fat mass with non-invasive methods (DEXA and RMN) will be assessed before and one-year after transplantation. Blood, before and after transplantation, as well as adipose tissue during transplantation surgery, will be sampled in order to constitute a blood, gene and tissue bank for defining the inflammatory status of this tissue using histological and molecular analysis.

Primary endpoint: The primary endpoint will be IL-7 blood levels in the different groups according to fat mass, metabolic parameters and immunosuppressive regimen. The hypothesis is that an increase of IL-7 levels, possibly induced by immunosuppressive regimen, is associated with quantitative and/or qualitative disturbances of adipose tissue and the development of insulin resistance.

Expected results and possible implications: This study will enable the consequences of immunosuppression on IL-7 levels, adipose tissue disturbances and glucose metabolism to be determined. Our approach combining clinical investigation and ex vivo and in vitro analysis is original and should result in better understanding of the cellular mechanisms responsible for the inflammatory process initiated in white adipose tissue and accompanying the disorders of this tissue (especially post-transplantation diabetes), thus opening new therapeutic perspectives in a major complication of transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* More than 18 years old
* BMI inferior to 30 kg/m2
* non diabetic patients who need a kidney or a liver transplantation(Glucose blood level <1,26 g/L without any antidiabetic drug)
* OR included in the islet transplantation protocol because of a C peptide negative brittle or difficult to treat diabetes.
* cover under the social security

Exclusion Criteria:

* Unable to receive enlightened information
* Refusal to sign the consent
* Auto immune disease (kidney, liver or chronic inflammatory disease)
* need for a kidney-pancreas transplantation
* Creatinin > 15 mg / L for patients non concerned by kidney transplantation
* Sepsis
* Oestrogens, raloxifene
* Active alcohol Intoxication
* Cancers or autoimmune diseases;
* Psychiatric Pathology
* Active infection including hepatitis C or HIV;
* Age under 18 years or above 65 years
* Participation in another study excluded the possibility of participating in another protocol
* No cover under the social security
* Pregnant or lactating women
* patients under guardianship, persons deprived of liberty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a transplantation in Endocrinology Metabolism department, Nephrology department and Liver Transplantation department in Lille University Hospital, Amiens University Hospital, Caen University Hospital, Rouen University Hospital and Reims University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
interleukin 7 | 1 year

SECONDARY OUTCOMES:
Interleukin 2 | 1 year
Interleukin 4 | 1 year
Interleukin 9 | 1 year
Interleukin 15 | 1year
Interleukin 21 | 1year
TNFa | 1 year
Interleukin 1b | 1 year
Interleukin 6 | 1year
Interleukin 8 | 1 year
Interleukin 10 | 1 year
Interleukin 18 | 1 year
leptin | 1 year
adiponectin | 1 year
Blood cells of innate and adaptative immunity analysis | 1 year
fat mass | 1 year
metabolic parameters | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine VANTYGHEM, MD, PhD, Principal Investigator — Lille University Hospital
Locations (5):
- France (5):
  - Amiens University Hospital, Amiens
  - Caen University Hospital, Caen
  - Lille University Hospital, Lille
  - Reims University Hospital, Reims
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No